CLINICAL TRIAL: NCT00973063
Title: Influence of Routine Sterile Gloving on Contamination Rates in Blood Culture
Brief Title: Effectiveness of Routine Sterile Gloving in Blood Culture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wan Beom Park, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0906-029-283; SNUHIMI01
Record Dates: First submitted 2009-09-07; First posted 2009-09-09 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: Bacteremia
Keywords: bacteremia; blood culture; contamination
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional gloving (No Intervention)
- routine sterile gloving (Experimental)
  Interventions: Behavioral: Routine sterile gloving

INTERVENTIONS:
Behavioral: Routine sterile gloving — routinely new sterile gloving just before sampling
  Arms: routine sterile gloving

SUMMARY:
The purpose of this study is to determine whether routine sterile gloving can lower contamination rates in blood culture.

DETAILED DESCRIPTION:
Because contamination during sampling for blood culture may interfere in interpreting the results of blood culture, lowering the contamination rates in blood culture is very important. According to current guideline, routine sterile gloving is not recommended. We hypothesized that routine sterile gloving can lower contamination rates in blood culture.

ELIGIBILITY:
Inclusion Criteria:

* The patients in whom Blood culture is medically needed

Exclusion Criteria:

* Blood sample is obtained through central venous catheter or arterial line
* No consent to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1854 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
contamination rate in blood culture | at the time of identification of organisms

CONTACTS AND LOCATIONS:
Overall Officials: WAN BEOM PARK, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim NH, Kim M, Lee S, Yun NR, Kim KH, Park SW, Kim HB, Kim NJ, Kim EC, Park WB, Oh MD. Effect of routine sterile gloving on contamination rates in blood culture: a cluster randomized trial. Ann Intern Med. 2011 Feb 1;154(3):145-51. doi: 10.7326/0003-4819-154-3-201102010-00003. PMID 21282693